CLINICAL TRIAL: NCT00756522
Title: Specialized Center of Clinically Oriented Research: Alveolar and Airway Mechanisms for COPD. Detection: Lung Imaging and Profiling (Project 1)
Brief Title: Analyzing Lung Tissue in People With and Without Chronic Obstructive Pulmonary Disease Who Are Undergoing Lung Transplantation
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 575-201109012
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, isolated RNA and DNA, and lung tissue
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: There is no intervention. Study is observational. — There is no intervention. Study is observational.

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a long-term lung disease. People with COPD have difficulty breathing because of lung damage. However, for many people with COPD, while some areas of the lungs are damaged, other nearby areas are not. This study will examine lung tissue from people with and without COPD who are undergoing lung transplantation to investigate how and why certain areas of the lungs are damaged in some people but not others.

DETAILED DESCRIPTION:
COPD is a common lung disease and is the fourth most common cause of death in the United States. Symptoms include coughing, excess mucus production, shortness of breath,and wheezing. There is no cure for COPD, and the disease worsens over time. Treatment can include stopping smoking, taking medications, receiving supplemental oxygen, and in severe cases, undergoing lung transplantation. COPD is usually the result of many years of cigarette smoking, but it remains unknown exactly how cigarette smoking causes this disease.

One reason that people with COPD experience shortness of breath and cough is because the lung airways are partly damaged and obstructed. In healthy people, oxygen is breathed in and then passes easily into the bloodstream through bunches of small air sacs that fill the lungs. In people with COPD, these air sacs are damaged, making it difficult for oxygen to pass into the bloodstream. However, even in people with severe COPD, the air sacs in some areas of the lungs continue to work, even though neighboring air sacs are damaged. It is possible that an overactive immune response may cause the air sac damage and that some people with COPD are more prone than others to such immune system abnormalities. By examining the differences in lung tissue in people with and without COPD who are undergoing a lung transplant, this study will investigate why some people's immune systems cause lung damage and others do not and how and why some air sacs are damaged while other nearby air sacs are not. Study researchers will also examine whether genetic factors play a role in the development and severity of COPD.

This study will enroll people with COPD who are undergoing lung transplantation. Before the lung transplantation surgery, participants will attend one study visit, which will include a medical history review, height and weight measurements, and a blood collection. A portion of blood will be stored for future genetic research. Participants will also complete questionnaires to collect information on activities, health, and quality of life. Some participants will undergo a 3-Helium magnetic resonance imaging (MRI) procedure, which is an imaging technique that allows doctors to see the air spaces inside of the lungs. After the lung transplantation surgery, study researchers will collect lung tissue from surgery. Study researchers will contact participants at the end of the study to collect follow-up medical information.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Ability to read and write in English
* Able to participate in the informed consent process
* Listed at Barnes-Jewish Hospital for lung transplantation for COPD (with alpha-1-antitrypsin deficiency [A1ATD] or non-1ATD)
* Global Initiative for Chronic Obstructive Lung Disease (GOLD) class IV COPD
* Acceptable chest computed tomography (CT) exam completed at Barnes-Jewish Hospital in the 3 years before study entry

Exclusion Criteria:

* Pregnant
* Prisoner
* Vulnerable populations
* Coexisting active chronic inflammatory or collagen vascular disease, immunodeficiency of any kind, non-cutaneous malignancy (melanoma is an exclusion), or previous organ transplant
* Coexisting (other than COPD / emphysema / chronic bronchitis)significant pulmonary parenchymal disorder (e.g., pulmonary fibrosis)

Exclusion Criteria for 3-Helium MRI Procedure:

* Inability to perform 10 to 15 second breath hold for 3-Helium MRI scan.
* Contraindications to MRI (including pacemaker, metal implants, other devices affected by the magnet).
* Contraindications to 3-Helium MRI (including significant anemia [hemoglobin less than or equal to 12 g/dL, with the last testing within 1 month of the MRI scan] or marked oxyhemoglobin desaturation at rest when breathing room air [requiring more than 4 liters per minute of supplemental oxygen to keep saturation of oxygen (SaO2) at least 90%]).However, patients deemed to be low risk kfor complications of cerebrovascular disease, cardiovascular disease, heart dysrhythmias, and seizures through the thorough lung transplant evaluation will be eligible for testing. Since most of the patients with these contraindications to 3-Helium MRI will be ineligible for lung transplantation, we expect few patients to have such contraindications to testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be adults with a clinically established need for lung transplantation and who are listed at Barnes-Jewish Hospital for lung transplantation because of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Pierce, PhD, Principal Investigator — Washington University School of Medicine, Pulmonary and Critical Care Division; Michael Holtzman, MD, Study Chair — Washington University School of Medicine, Pulmonary and Critical Care Division
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States